CLINICAL TRIAL: NCT06203223
Title: The Effect of Ovamax on Oocyte Quality in Women Undergoing IVF
Brief Title: The Effect of Ovamax on Oocyte Quality
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was stopped prematurely due to low recruitment rate
Sponsor: Aristotle University Of Thessaloniki (Other)
Collaborators: Eugonia IVF Unit, Athens, Greece (Other)
Responsible Party: Principal Investigator, E.M. Kolibianakis, Professor of Obstetrics Gynaecology and Assisted Reproduction, Aristotle University Of Thessaloniki
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UHR-17
Record Dates: First submitted 2022-01-11; First posted 2024-01-12 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Female; Infertility
Keywords: oocyte quality assessment; oocyte scoring; antioxidants; ivf
MeSH Terms: conditions — Infertility; Long Qt Syndrome 3

STUDY DESIGN:
Intervention Model Description: randomised controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: use of placebo, masked randomisation list
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ova-max (Active Comparator): antioxidant, dietary supplement
  Interventions: Other: Ova-max
- Placebo (Placebo Comparator): placebo
  Interventions: Other: placebo

INTERVENTIONS:
Other: Ova-max — use Ova-max 3 months prior to treatment initiation
  Arms: Ova-max
Other: placebo — use placebo 3 months prior to treatment initiation
  Arms: Placebo

SUMMARY:
Oocyte quality is a basic parameter that affects embryo quality and therefore it influences the outcome of assisted reproduction. It has been suggested that oocyte quality is improved by the intake of vitamins and antioxidants.

Ova-Max is a dietary supplement that consists of vitamins, minerals and antioxidants which improve women's oocytes by preventing oxidative stress. Specifically, Ovamax includes Chasteberry, Melatonin, Myo-Inositol, Folic Acid, Co-Enzyme Q10, Vitamin E, L-Arginine, Grape seed extract and Alpha-lipoic Acid. The purpose of this study is to evaluate the influence of Ova-max intake on oocyte quality in women undergoing In Vitro Fertilization.

According to the research hypothesis the administration of Ova-Max for three months increases oocyte quality in women undergoing intracellular sperm injection after ovarian stimulation and oocyte retrieval.

DETAILED DESCRIPTION:
Randomisation

This study is a blind randomized control trial to evaluate the association between Ova-Max intake and the quality of oocytes retrieved after ovarian stimulation. Randomization will be performed at least three months prior to initiation of treatment and patients will be assigned to either Ova-max or placebo by a computer-generated randomization list.

Ovarian Stimulation

A standard ovarian stimulation protocol for all patients will be followed with 200-300 IU of recombinant FSH and GnRH antagonist starting on day 5 of stimulation.

Induction of final oocyte maturation will be performed by recombinant hCG or GnRH agonist. Women who are planned for fresh embryo transfer, will be administered subcutaneous progesterone for luteal phase support starting on the day of oocyte retrieval.

Oocyte Quality Assessment

After oocyte retrieval the cumulus cells of the Cumulus Oocyte complex (COC) are removed and quality of all mature, metaphase II (MII) oocytes is assessed according to the following parameters:

1. Oocyte shape
2. Oocyte size
3. Ooplasm characteristics
4. Structure of the perivitelline space (PVS)
5. Zona pellucida (ZP) and
6. Polar body (PB) morphology

Each parameter is graded as worst (-1), average (0), or best (1) and a total oocyte score (TOS) is calculated by summing up individual parameter assessments.

The maximal TOS of an oocyte, therefore, could be +6, the lowest -6.

The 6 individual parameters are assessed in detail as follows:

1. Oocyte shape (-1): poor oocyte morphology (dark general oocyte coloration and/or ovoid shape) (0): almost normal (less dark general oocyte coloration and less ovoid shape) (+1): normal
2. Oocyte size (-1): abnormally small or large oocyte (0): almost normal size (+1): oocyte size was within normal range
3. Ooplasm characteristics (-1): very granulated and/or very vacuolated cytoplasm and/or demonstrated several inclusions (0): slightly granular and/or demonstrated only few inclusions (+1): absence of granularity and inclusions
4. Structure of the perivitelline space (PVS) (-1): abnormally large PVS, absence of PVS or very granular PVS (0): moderately enlarged PVS and/or small PVS and/or a less granular PVS (+1): normal size PVS with no granules
5. Zona pellucida (ZP) (-1): very thin or thick ZP (0): small deviation from normal (+1): normal zona
6. PB morphology (+1): flat and/or multiple PBs, granular and/or either abnormally small or large PB (0): fair but not excellent PB (+1): normal size and shape of PB

After having assessed the TOS of all MII oocytes, the Mean Oocyte Score (MOS) of the patient is calculated by dividing the sum of all TOS of the patient by the number of her oocytes.

Statistical analysis

Group sample sizes of 79 and 79 achieve 80% power to detect a difference of -1.0 between the null hypothesis that both group TOS means are -1.1 and the alternative hypothesis that the mean TOS of the Ova-Max group is -0.1, with known group standard deviations of 2.2 and 2.2 and with a significance level (alpha) of 0.05000 using a two-sided Mann-Whitney test assuming that the actual distribution is uniform

ELIGIBILITY:
Inclusion Criteria:

* Patients less than 46 years of age
* ICSI for fertilisation to allow evaluation of oocyte quality

Exclusion criteria:

* Women with endometriosis
* Women with only one ovary
* More than two previous IVF cycles
* Use of testicular sperm
* Intake of other dietary supplements
* Poor responders

Ages: 18 Years to 46 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 97 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2025-01-15 (Actual)

PRIMARY OUTCOMES:
Mean oocyte score | 1-3 hours after oocyte retrieval
  The sum of the total oocyte scores of the patient divided by the number of her oocytes.
  Oocytes is assessed according to the following parameters:
  1. Oocyte shape
  2. Oocyte size
  3. Ooplasm characteristics
  4. Structure of the perivitelline space (PVS)
  5. Zona pellucida (ZP) and
  6. Polar body (PB) morphology
  Each parameter is graded as worst (-1), average (0), or best (1) and a total oocyte score (TOS) is calculated by summing up individual parameter assessments.
  The maximal TOS of an oocyte, therefore, could be +6, the lowest -6.

SECONDARY OUTCOMES:
Percentage of mature oocytes | 2-4 hours after oocyte retrieval
  number of mature oocytes of a woman divided by her total oocyte number
Percentage of fertilised oocytes | 16-18 hours after fertilisation
  number of oocytes of a woman that are fertilised divided by the total oocyte injected with sperm
Blastulation rate | day 5 after fertilisation
  the number of embryos that have reached blastocyst stage divided by the number of fertilised oocytes
Pregnancy rate | 6 weeks after embryo transfer
  the number of women who got pregnant divided by the number of women who underwent embryo transfer
Total number of COCs collected | immediately after oocyte retrieval
  total number of cumulus oocyte complexes collected from each woman

CONTACTS AND LOCATIONS:
Overall Officials: Efstratios M Kolibianakis, Professor, Principal Investigator — Aristotle University Thessaloniki
Locations (1):
- Papageorgiou Hospital, Thessaloniki, Central Macedonia, Greece

IPD SHARING:
Plan to Share IPD: No